CLINICAL TRIAL: NCT05935085
Title: A Phase 2, Randomized, Double Blind, Placebo Controlled Study to Evaluate the Efficacy and Safety of ANB032 in the Treatment of Subjects with Moderate to Severe Atopic Dermatitis
Brief Title: This Study Will Evaluate the Safety, Tolerability, and Efficacy of ANB032 in Subjects with Moderate to Severe Atopic Dermatitis (AD).
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: ANB032 did not meet the primary endpoint in moderate-to-severe atopic dermatitis
Sponsor: AnaptysBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANB032-201
Record Dates: First submitted 2023-06-06; First posted 2023-07-07 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2024-08

CONDITIONS: Atopic Dermatitis Eczema
Keywords: ANB032, B and T lymphocyte attenuator BTLA

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- ANB032 SC Dose 1 (Experimental): This arm will receive treatment SC
  Interventions: Drug: ANB032
- ANB032 SC Dose 2 (Experimental): This arm will receive treatment SC
  Interventions: Drug: ANB032
- ANB032 SC Dose 3 (Experimental): This arm will receive treatment SC
  Interventions: Drug: ANB032
- Placebo (Placebo Comparator): This arm will receive Placebo SC
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ANB032 — BTLA agonist antibody
  Arms: ANB032 SC Dose 1; ANB032 SC Dose 2; ANB032 SC Dose 3
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study will evaluate the safety, tolerability, and efficacy of ANB032 in subjects with moderate to severe atopic dermatitis (AD).

DETAILED DESCRIPTION:
This is a Phase 2, randomized, double blind, placebo controlled, parallel group, multicenter study to evaluate the safety, tolerability, efficacy, pharmacokinetics, and immunogenicity of ANB032 in subjects with moderate to severe atopic dermatitis (AD).

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female aged 18 to 65 years and in good general health
* Moderate to severe AD for at least 6 months prior to Randomization
* History of inadequate response to treatment for AD with topical medications or for whom topical treatments are otherwise medically inadvisable
* EASI score ≥ 16 at Screening and at Randomization
* vIGA AD score ≥ 3 at Screening and at Randomization
* AD involved BSA ≥ 10% at Screening and at Randomization

Key Exclusion Criteria:

* Any factors that in the Investigator's opinion would predispose the subject to develop an infection
* Known or suspected congenital or acquired immunodeficiency state, or condition that would compromise the subject's immune status
* Not able to tolerate SC drug administration
* Tanning booth use or extended sun exposure that could affect disease severity or interfere with disease assessments within 4 weeks before Randomization

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2023-06-13 (Actual); Primary Completion 2024-10-16 (Actual); Study Completion 2025-01-07 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who achieve ≥75% reduction (improvement) from Baseline in EASI-75 as Week 14 | Baseline to Week 14
  The EASI is a validated measure used in clinical practice and clinical trials to assess the severity and extent of AD. The EASI is a composite index with scores ranging from 0 to 72.

SECONDARY OUTCOMES:
Mean percent change from Baseline in EASI at Week 14 | Baseline to Week 14
  The EASI is a validated measure used in clinical practice and clinical trials to assess the severity and extent of AD. The EASI is a composite index with scores ranging from 0 to 72.
Mean change from Baseline in EASI at Week 14 | Baseline to Week 14
Proportion of subjects who achieve a vIGA-AD score of 0 or 1 and ≥ 2-point reduction (improvement) from Baseline in vIGA-AD score at Week 14 | Baseline to Week 14

CONTACTS AND LOCATIONS:
Overall Officials: Mark Rigby, MD, Study Director — AnaptysBio, Inc.
Locations (78):
- United States (41):
  - AnaptysBio Investigative Site 10-140, Anaheim, California
  - AnaptysBio Investigative Site 10-141, Cerritos, California
  - AnaptysBio Investigative Site 10-121, Fountain Valley, California
  - AnaptysBio Investigative Site 10-107, Fremont, California
  - AnaptysBio Investigative Site 10-120, Lancaster, California
  - AnaptysBio Investigative 10-125, Lomita, California
  - AnaptysBio Investigative Site 10-146, Oxnard, California
  - AnaptysBio Investigative Site 10-147, Pasadena, California
  - AnaptysBio Investigative Site 10-112, Santa Monica, California
  - AnaptysBio Investigative Site 10-136, Doral, Florida
  - AnaptysBio Investigative Site 10-133, Miami, Florida
  - AnaptysBio Investigative Site 10-116, Miami, Florida
  - AnaptysBio Investigative Site 10-134, Miami, Florida
  - AnaptysBio Investigative Site 10-106, Miami, Florida
  - AnaptysBio Investigative Site 10-122, Atlanta, Georgia
  - AnaptysBio Investigative Site 10-130, Boise, Idaho
  - AnaptysBio Investigative Site 10-151, Flossmoor, Illinois
  - AnaptysBio Investigative Site 10-127, Clarksville, Indiana
  - AnaptysBio Investigative Site 10-149, Merrillville, Indiana
  - AnaptysBio Investigative Site 10-128, New Albany, Indiana
  - AnaptysBio Investigative Site 10-137, Baton Rouge, Louisiana
  - AnaptysBio Investigative Site 10-131, Methuen, Massachusetts
  - AnaptysBio Investigative Site 10-126, Ann Arbor, Michigan
  - AnaptysBio Investigative Site 10-139, Auburn Hills, Michigan
  - AnaptysBio Investigative Site 10-114, Detroit, Michigan
  - AnaptysBio Investigative Site 10-138, Troy, Michigan
  - AnaptysBio Investigative Site 10-150, Hazelwood, Missouri
  - AnaptysBio Investigative Site 10-110, Saint Joseph, Missouri
  - AnaptysBio Investigative Site 10-148, Las Vegas, Nevada
  - AnaptysBio Investigative Site 10-109, Charlotte, North Carolina
  - AnaptysBio Investigative Site 10-108, Wilmington, North Carolina
  - AnaptysBio Investigative Site 10-129, Mason, Ohio
  - AnaptysBio Investigative Site 10-113, Portland, Oregon
  - AnaptysBio Investigative Site 10-145, Philadelphia, Pennsylvania
  - AnaptysBio Investigative Site 10-119, Nashville, Tennessee
  - AnaptysBio Investigative Site 10-144, Baytown, Texas
  - AnaptysBio Investigative Site 10-124, Dallas, Texas
  - AnaptysBio Investigative Site 10-105, Frisco, Texas
  - AnaptysBio Investigative Site 10-142, Katy, Texas
  - AnaptysBio Investigative Site 10-104, San Antonio, Texas
  - AnaptysBio Investigative Site 10-132, Spokane, Washington
- Australia (2):
  - AnaptysBio Investigative Site 35-103, Woolloongabba, Queensland
  - AnaptysBio Investigative Site 35-104, Coorparoo
- Canada (6):
  - AnaptysBio Investigative Site 11-105, Surrey, British Colombia
  - AnaptysBio Investigative Site 11-102, Barrie, Ontario
  - AnaptysBio Investigative Site 11-106, Etobicoke, Ontario
  - AnaptysBio Investigative Site 11-101, London, Ontario
  - AnaptysBio Investigative Site 11-103, North Bay, Ontario
  - AnaptysBio Investigative Site 11-107, Richmond Hill, Ontario
- Czechia (4):
  - AnaptysBio Investigative Site 57-104, Pardubice
  - AnaptysBio Investigative Site 57-105, Prague
  - AnaptysBio Investigative Site 57-102, Prague
  - AnaptysBio Investigative Site 57-101, Prague
- Georgia (7):
  - AnaptysBio Investigative Site 59-105, Tbilisi
  - AnaptysBio Investigative Site 59-106, Tbilisi
  - AnaptysBio Investigative Site 59-101, Tbilisi
  - AnaptysBio Investigative Site 59-102, Tbilisi
  - AnaptysBio Investigative Site 59-103, Tbilisi
  - AnaptysBio Investigative Site 59-104, Tbilisi
  - AnaptysBio Investigative Site 59-107, Tbilisi
- New Zealand (4):
  - AnaptysBio Investigative Site 36-101, Grafton
  - AnaptysBio Investigative Site 36-104, Nelson
  - AnaptysBio Investigative Site 36-102, Rosedale
  - AnaptysBio Investigative Site 36-103, Wellington
- Poland (14):
  - AnaptysBio Investigative Site 30-111, Bydgoszcz
  - AnaptysBio Investigative Site 30-113, Częstochowa
  - AnaptysBio Investigative Site 30-108, Gdansk
  - AnaptysBio Investigative Site 30-106, Krakow
  - AnaptysBio Investigative Site 30-101, Lodz
  - AnaptysBio Investigative Site 30-109, Rzeszów
  - AnaptysBio Investigative Site 30-115, Skierniewice
  - AnaptysBio Investigative Site 30-112, Szczecin
  - AnaptysBio Investigative Site 30-102, Świdnik
  - AnaptysBio Investigative Site 30-105, Warsaw
  - AnaptysBio Investigative Site 30-107, Warsaw
  - AnaptysBio Investigative Site 30-116, Warsaw
  - AnaptysBio Investigative Site 30-104, Wroclaw
  - AnaptysBio Investigative Site 30-114, Wroclaw

IPD SHARING:
Plan to Share IPD: No